CLINICAL TRIAL: NCT00725985
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Trial of Oral Cladribine in Subjects With a First Clinical Event at High Risk of Converting to MS
Brief Title: Oral Cladribine in Early Multiple Sclerosis (MS)
Acronym: ORACLE MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28821
Record Dates: First submitted 2008-07-30; First posted 2008-07-31 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome (CIS); Early MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Cladribine 5.25 mg/kg (ITP) (Experimental): Cladribine tablets administered as cumulative dose of 0.875 mg/kg over a course of 5 consecutive days at Weeks 1, 5, 9, 13, 48, and 52 resulting in total cladribine dose of 5.25 milligrams per kilograms (mg/kg) during the ITP of 96 weeks or until clinically definite multiple sclerosis (CDMS) conversion, whichever occurred first.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Cladribine 3.5 mg/kg (ITP) (Experimental): Cladribine tablets administered as cumulative dose of 0.875 mg/kg over a course of 5 consecutive days at Weeks 1, 5, 48, 52 and placebo matched to cladribine tablets was administered at Week 9 and 13 resulting in total cladribine dose of 3.5 mg/kg during the ITP of 96 weeks or until CDMS conversion, whichever occurred first.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Placebo (ITP) (Placebo Comparator): Placebo matched to cladribine tablets administered over a course of 5 consecutive days at Weeks 1, 5, 9, 13, 48 and 52 during the ITP of 96 weeks or until CDMS conversion, whichever occurred first.
  Interventions: Drug: Placebo; Drug: Rebif® new formulation (RNF)
- Cladribine 5.25 mg/kg, Rebif (OLMP) (Experimental): Participants who received cladribine 5.25 mg/kg and converted to CDMS during ITP entered in open-label maintenance period (OLMP) and received Rebif® new formulation (RNF) subcutaneously at a dose of 44 microgram (mcg) three times a week for up to 96 weeks. Due to trial termination, the OLMP duration was reduced for some participants.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Cladribine 3.5 mg/kg, Rebif (OLMP) (Experimental): Participants who received cladribine 3.5 mg/kg and converted to CDMS during ITP entered in OLMP and received RNF subcutaneously at a dose of 44 mcg three times a week for up to 96 weeks. Due to trial termination, the OLMP duration was reduced for some participants.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Placebo, Rebif (OLMP) (Experimental): Participants who received placebo and converted to CDMS during ITP entered in OLMP and received RNF subcutaneously at a dose of 44 mcg three times a week for up to 96 weeks. Due to trial termination, the OLMP duration was reduced for some participants.
  Interventions: Drug: Placebo
- Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (Experimental): Participants who received cladribine 5.25 mg/kg and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (Experimental): Participants who received cladribine 3.5 mg/kg and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) (Experimental): Participants who received placebo and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Placebo
- Cladribine 5.25 mg/kg, Rebif (LTFU) (Experimental): Participants who received cladribine 5.25 mg/kg and did not convert to CDMS during ITP, entered in LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU period received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Cladribine 3.5 mg/kg, Rebif (LTFU) (Experimental): Participants who received cladribine 3.5 mg/kg and did not convert to CDMS during ITP, entered in LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU period received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Cladribine; Drug: Rebif® new formulation (RNF)
- Placebo, Rebif (LTFU) (Experimental): Participants who received placebo and did not convert to CDMS during ITP, entered in LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who convert to CDMS during LTFU period received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cladribine — Cladribine tablets were administered until CDMS conversion, whichever occur first.
  Arms: Cladribine 3.5 mg/kg (ITP); Cladribine 3.5 mg/kg, Rebif (LTFU); Cladribine 3.5 mg/kg, Rebif (OLMP); Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU); Cladribine 5.25 mg/kg (ITP); Cladribine 5.25 mg/kg, Rebif (LTFU); Cladribine 5.25 mg/kg, Rebif (OLMP); Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU)
Drug: Placebo — Placebo matched to cladribine tablets were administered.
  Arms: Placebo (ITP); Placebo, Rebif (LTFU); Placebo, Rebif (OLMP); Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Drug: Rebif® new formulation (RNF) — Participants who converted to CDMS during ITP entered in open-label maintenance period (OLMP) and received RNF subcutaneously at a dose of 44 microgram (mcg) three times a week. Participants who converted to CDMS during long-term follow-up (LTFU) period, received RNF subcutaneously at a dose of 44 mcg three times a week.
  Arms: Cladribine 3.5 mg/kg (ITP); Cladribine 3.5 mg/kg, Rebif (LTFU); Cladribine 3.5 mg/kg, Rebif (OLMP); Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU); Cladribine 5.25 mg/kg (ITP); Cladribine 5.25 mg/kg, Rebif (LTFU); Cladribine 5.25 mg/kg, Rebif (OLMP); Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU); Placebo (ITP)

SUMMARY:
A randomized, double-blind, clinical trial to assess the safety and efficacy of two doses of oral cladribine versus placebo in participants who had a first clinical demyelinating event (clinically isolated syndrome). Participants in either the cladribine or placebo group may also enter treatment periods with open-label interferon-beta or open-label cladribine depending upon the disease status. The primary objective of this study is to evaluate the effect of two dosage regimens of oral cladribine versus placebo on the time to conversion to multiple sclerosis (MS) (from randomization) according to the Poser criteria in participants with first clinical demyelinating event at high risk of converting to MS.

DETAILED DESCRIPTION:
This will be a randomized, double blind, three-arm, placebo-controlled, multi-center trial to evaluate the safety and efficacy of oral cladribine versus placebo in the treatment of participants who have sustained a first clinical demyelinating event within 75 days prior to the Screening. Participants must have a minimum of 2 clinically silent lesions on the Screening magnetic resonance imaging (MRI).

The study will include a pre-study evaluation period (Screening period: between 10 and 28 days prior to the start of treatment with blinded study medication (oral cladribine or placebo).

Depending upon the clinical course of their MS, participants will then proceed from the ITP to either the Maintenance Treatment Period (with open-label interferon-beta treatment) or LTFU period (with either open-label low-dose cladribine or no additional treatment (if no progression to MS has been noted after the initial treatment period). The single primary endpoint for the overall study, which will be determined during the ITP, is time to conversion to MS (from randomization), according to the Poser criteria.

For every participants, eligibility for study enrollment and entry into each of the study periods, and diagnosis of conversion to either McDonald MS or CDMS must be confirmed and approved by a Sponsor appointed study Adjudication Committee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years old, inclusive
* Weighed between 40 to 120 kilogram (kg), inclusive
* Participant has experienced a single, first clinical event suggestive of MS within 75 days prior to the Screening visit, (clock starts 24 hours after onset). The event must be a new neurological abnormality present for at least 24 hours, either mono- or polysymptomatic
* Participant has at least two clinically silent lesions on the T2-weighted MRI scan, at screening, with a size of at least 3 millimeter (mm), at least one of which is ovoid or periventricular or infratentorial on screening MRI
* Participant has EDSS 0 - 5.0 at Screening
* Participant has no medical history or evidence of latent tuberculosis infection (LTBI) or active tubercular disease, as evidenced by the Mantoux tuberculosis (TB) skin test or a comparable sensitive test according to local regulations/guidelines (if the Mantoux test is not available), and/or a chest X-ray
* Participant has normal hematological parameters at Screening, as defined by the central laboratory that performed all the assessments
* If female, she must:

  * be neither pregnant nor breast-feeding, nor attempting to conceive and
  * use a highly effective method of contraception throughout the entire duration of the study and for 90 days following completion of the last dose of study medication. A highly effective method of contraception is defined as those which result in a low failure rate (that is less than 1 percent per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner, or
  * be post-menopausal or surgically sterilized (Note: for Danish sites only, participants should use a hormonal contraceptive or intrauterine device for the duration of the trial)
* Male participants must be willing to use contraception to avoid impregnating partners throughout the study, and for 90 days following the last dose of study medication
* Be willing and able to comply with study procedures for the duration of the study
* Participant has to provide written informed consent voluntarily, including, for United states of America (USA), participant authorization under Health Insurance Portability and Accountability Act (HIPAA), prior to any study-related procedure that is not part of normal medical care
* Participant has refused any treatment already available for clinically isolated syndrome (CIS) such as interferons or glatiramer acetate, at the time of entry into the Initial Treatment Period of this study

Exclusion Criteria:

* Participant has a diagnosis of MS (per McDonald criteria, 2005)
* Participant has any other disease that could better explain the participant's signs and symptoms
* Participant has complete transverse myelitis or bilateral optic neuritis
* Participant using or has used any other approved MS disease modifying drug (DMD)
* Participant has used any investigational drug or undergone an experimental procedure within 12 weeks prior to Study day 1
* Participant received oral or systemic corticosteroids or adrenocorticotropic hormone (ACTH) within 30 days prior to screening MRI. The MRI had to be performed 30 days after the oral or systemic corticosteroids or ACTH treatment. In case this interfered with MRI timing the screening period could be extended accordingly.
* Participant has abnormal total bilirubin, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase greater than 2.5 times the upper limit of normal
* Participant suffered from current autoimmune disease other than MS
* Participant suffered from psychiatric illness (including history of, or concurrent, severe depressive disorders and/or suicidal ideation) that in the opinion of the investigator creates undue risk to the participant or could affect compliance with the study protocol
* Participant suffered from major medical illness such as cardiac (for example angina, congestive heart failure or arrhythmia), endocrinologic, hepatic, immunologic, metabolic, renal, pulmonary, gastrointestinal, dermatologic, or other major disease that would preclude the administration of oral cladribine
* Participant has a history of seizures not adequately controlled by medications
* Participant has a known allergy to cladribine, interferon-beta, the excipient(s) of the study medications, or to gadolinium- diethylenetriamine penta-acetic acid (DTPA)
* Participant has any renal condition that would preclude the administration of gadolinium (for example acute or chronic severe renal insufficiency (glomerular filtration rate [GFR] less than 30 milliliter per minute per 1.73 square meter [mL/min/1.73 m^2])
* Participant has a history of chronic or clinically significant hematological abnormalities
* Participant has a history of active or chronic infectious disease or any disease that compromises immune function (for example human immunodeficiency virus positive [HIV+], human T-lymphotrophic virus [HTLV-1], Lyme disease, latent tuberculosis infection [LTBI] or TB, insulin-dependent diabetes).
* Participant has previously been screened in this study (signed an informed consent) and then withdrawn
* Participant has received any immunomodulatory or immunosuppressive therapy) at any time prior to Study Day 1, including, but not limited to, the following products: any interferon, glatiramer acetate (Copolymer I), cyclophosphamide, cyclosporine, methotrexate, linomide, azathioprine, mitoxantrone, teriflunomide, laquinimod, cladribine, total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment (for example natalizumab, alemtuzumab/Campath, anti-cluster of differentiation 4 [CD4]), intravenous immunoglobulin G (IVIG), cytokines or anti-cytokine therapy
* Participant has received experimental MS treatment
* Participant has a history of alcohol or drug abuse
* Participant has intolerance or any contraindication to both paracetamol (acetaminophen) and ibuprofen
* Participant has inability to administer subcutaneous injections either by self or by caregiver
* Participant has prior or current malignancy (with the exception of in situ basal or squamous cell skin cancer surgically removed without recurrence for at least five years)
* Participant has a positive stool hemoccult test at Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 617 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2012-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Stubinski, MD, Study Director — Merck Serono S.A., Geneva
Locations (158):
- United States (24):
  - Hope Research Institute Medical Plaza LLC Desert Hills, Phoenix, Arizona
  - Multiple Sclerosis Center Drive, Neurology Suite 701, Newport Beach, California
  - University of Colorado at Denver Health Sciences, Denver, Colorado
  - Fort Collins Neurology, Fort Collins, Colorado
  - MS Center of Brevard MIMA Centry Research Associates, Melbourne, Florida
  - University of South Florida, Tampa, Florida
  - MS Center of Atlanta, Atlanta, Georgia
  - Bruce Hughes West Building, Des Moines, Iowa
  - Michigan Neurology Associates, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Dennis Dietrich, Great Falls, Montana
  - University of Medicine and Dentistry of New Jersey School of Neurology, Stratford, New Jersey
  - Upstate Clinical Research LLC 3, Albany, New York
  - Neurological Specialists of Long Island, Great Neck, New York
  - Multiple Sclerosis Center of Northeastern NY, New York, New York
  - Comprehensive MS Care Clinic at South Shore Multiple Sclerosis, Patchogue, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Meritcare Neuroscience Center Neurology, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - MS Center of Oklahoma, Oklahoma City, Oklahoma
  - Neurology and Sleep Medicine, Bethlehem, Pennsylvania
  - Swedish Medical Center Cherry Hill, Seattle, Washington
  - Neurology & Neurological Association of Tacoma, Tacoma, Washington
- Argentina (2):
  - Instituto Medico Rodriguez Alfici, Godoy Cruz
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
- Krankenhaus der Barmherzigen Brüder, Linz, Austria
- Belgium (4):
  - Algemeen Ziekenhuis St Jan, Bruges
  - Cliniques Universitaires St-Luc, Brussels
  - Hopital Erasme, Brussels
  - CHU de Liege - Domaine Universitaire du Sart Tilman,, Liège
- Clinical Center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (9):
  - Military Medical Academy- Sofia (MMA), Pleven
  - MBAL Rousse AD 1st, Rousse
  - Central Clinic Hospital, Sofia
  - Military Medical Academy, Sofia
  - National Heart Hospital, Sofia
  - Second MHAT, Sofia
  - Tokuda Hospital, Sofia
  - University Hospital St Naum, Sofia
  - Medical Centre Centromed 2000, Veliko Tarnovo
- Ottawa General Hospital, Ottawa, Canada
- Croatia (2):
  - General Hospital Varazdin, Varaždin
  - University Hospital Zagreb, Zagreb
- Czechia (6):
  - Faculty Hospital Brno, Brno
  - Neurological dept of Faculty, Hradec Králové
  - Fakultní nemocnice s poliklinikou Ostrava, Ostrava
  - Faculty Hospital Motol, Prague
  - Klinika Vseobecne, Prague
  - Nemocnice Teplice, Teplice
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
- Finland (5):
  - HUS Hyvinkaa Central Hospital, Hyvinkää
  - OYKS Neurologian Klinikka, Oulu
  - Neurologian Klinikka Seinajoen Keskussairaala, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turun Yliopistollinen Keskussairaala Rakennus 3 1, Turku
- France (3):
  - CHU de Lille, Lille
  - CHU de Nantes, Nantes
  - American Memorial Hospital, Reims
- Georgia (3):
  - David Tatishvili Medical Center, Tbilisi
  - Medical Center Health, Tbilisi
  - S. Khechinashvili Tbilisi State Medical University, Tbilisi
- Germany (2):
  - Universitaetsklinikum und Medizinische Fakultaet Heidelberg, Heidelberg
  - Philipps-Universitaet Marburg, Marburg
- India (6):
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - St.John's Medical College and Hospital, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences and Research, Kochi, Kerala
  - Kovai Medical Centre and Hospital, Coimbatore
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Mallikatta Neuro and Research Centre, Mangalore
- Italy (17):
  - Ospedale Regionale Torrette, Ancona
  - Università de Bari, Bari
  - Ospedale Binaghi Centro Sclerosi Multipla, Cagliari
  - Azienda Ospedaliera Garibaldi, Catania
  - Dipartimento di Neuroscienze, Catania
  - Università G. D'Annunzio, Chieti
  - Ospedale San Antonio Abate, Gallarate
  - Universita degli Studi di Genova, Genova
  - Ospedale e casa di riposo P. Richiedei, Gussago
  - Ospedale San Raffaele, Milan
  - Dipartimento di Scienze Neurologiche, Napoli
  - Azienda Sanitaria Ospedaliera San Luigi Gonzaga, Orbassano
  - Villa Sofia Hospital Azienda Ospedaliera Villa Sofia P.zza Salerno e Resuttana 1, Palermo
  - Istituto Neurologico C. Mondino, Pavia
  - Azienda Ospedaliera S. Camillo Forlanini, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Università di Roma La Sapienza, Roma
- American University of Beirut, Beirut, Lebanon
- Clinic of Neurology "Klinicki Centar", Skopje, North Macedonia
- Norway (2):
  - Helse Bergen HF Kvinneklinikken Haukeland Universitetssykehus Jonas, Bergen
  - Regionsykehuset I Trondheim, Nevrologisk avd., Trondheim
- Poland (9):
  - 10 Wojskowy Szpital Kliniczny, Bydgoszcz
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Gdansk
  - Niepubliczny Zespol Opieki Zdrowotnej, Krakow
  - Medical Academy of Lodz, Lodz
  - Panstwowy Szpital Kliniczny, Lublin
  - Wojewodzki Szpital Specjalistyczny Oddział Neurologii z Pododdziałem Udarowym, Olsztyn
  - Medical Academy, Poznan
  - Medical Academy II, Warsaw
  - Medical Academy, Warsaw
- Portugal (4):
  - Hospital Fernando da Fonseca, Amadora
  - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de Coimbra, S. Martinho Do Bispo
- Romania (4):
  - "Dr. Carol Davilla" Military Clinical Hospital, Bucharest
  - Centrul Medical SANA, Bucharest
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - County Hospital Timisoara, Timișoara
- Russia (25):
  - Municipal Healthcare Institution "City Clinical Hospital #3", Chelyabinsk
  - State Healthcare Institution "Kaluga Regional Hospital", Kaluga
  - State Medical Institution "Republican Rehabilitation Clinic of Tatarstan Ministry of Health", Kazan'
  - State Healthcare Institution "Kemerovo Regional Clinical Hospital", Kemerovo
  - State Medical Institution " Jursk Regional Clinical Hospital", Kursk
  - Moscow State Healthcare Institution City Clinical Hospital #11, Moscow
  - Non-State Healthcare Institution "Central Clinical Hospital #2 named after N.A. Semasko of Russian Railways", Moscow
  - State Educational Institute of Higher Professional Education "I.M. Sechenov Moscow Medical Academy of Roszdrav" Russia based on A. Ya. Kozhevnikov Nervous Disease Clinic, Moscow
  - Municipal Treatment Prophylactic Institution "City Hospital #33", Nizhny Novgorod
  - Federal State Institution " Siberian Reginal Medical Center of Roszdarv", Novosibirsk
  - State institution Science Research Institute Clinical and Experimental Lymphology of Russian Academy of Medical Sciences, Novosibirsk
  - State Educational Institute of Higher Professional Education "Rostov State Medical University of Roszdrav", Rostov-on-Don
  - State Healthcare Institution "Rostov Region Clinical Hospital", Rostov-on-Don
  - Institute of Human Brain of Russian Academy of Science Dept. of Multiple Sclerosis, Saint Petersburg
  - International Clinic and Hospital, Neurology, Saint Petersburg
  - St. Petersburg State Healthcare Institution "Multifield City Hospital #2", Saint Petersburg
  - State Educational Institution of Higher Professional Education "Military Medical Academy named after S. M. Korov of Dept of Defense of Russian Federation based on Clinic of Neurology of State Institution, Saint Petersburg
  - State Educational Institution of Higher Professional Education "Samara State Medical University of Roszdrav" on State Healthcare Institution "Samara Regional Clinical Hospital named after M. I. Kalinin", Samara
  - State Educational Institution of Higher Professional Education "Saratov State Medical University of Roszdrav" based on Clincial Hosptial #3 of Saratov State Medical University, Saratov
  - Regional State Healthcare Institution "State Smolensk Region Clinical Hospital", Smolensk
  - State Educational Institution of Higher Professional Education "Siberian State Medical University of Roszdrav", Tomsk
  - Closed joint-stock society Medical sanitary unit "Nephtaynik" based the hospital, Tyumen
  - Vladimir Regional State Healthcare Institution "Regional Clinical Hospital", Vladimir
  - Municipal Healthcare Institution "Yaroslavi Clinical Hospital #8", Yaroslavl
  - State Healthcare Institution "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg
- Serbia (3):
  - Clinical Centre of Serbia, Belgrade
  - Hospital for Prevention and Treatment of Cerebro-Vascular Diseases, Belgrade
  - Clinical Centre Niš, Niš
- National Neuroscience Institute (TTSH Campus), Singapore, Singapore
- South Korea (5):
  - National Cancer Center, Department of Neurology,, Gyeonggi-do
  - Department of Neurology, 50 Ilwon-dong, Gangnam-gu, Seoul
  - Department of Neurology, Asan Medical Center, 388-1 Pungnap 2-dong, Songpa-gu, Seoul
  - Seoul National University Hospital, Department of Neurology, Seoul
  - Yonsei University Medical Center, Department of Neurology, Yonsei University Medical Center, Seoul
- Spain (2):
  - Hospital Reina Sofia Cordoba, Córdoba
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz de Tenerife
- Sweden (3):
  - Sahlgrenskasjukhuset, Gothenburg
  - Karolinska University Hospital, Stockholm
  - Umea University Hospital, Umeå
- Taiwan (2):
  - Taipei Veterans, Taipei
  - Chang Gung Medical Foundation- Linkou Branch No5, Taoyuan District
- Srinagarind Hospital, Khon Kaen, Thailand
- Turkey (Türkiye) (2):
  - Dokuz Eylul University, Izmir
  - Ondokuz Mayis Universitesi, Samsun
- Ukraine (3):
  - State Established "Institute of Neurology, Psychiatry and Narcology of the AMS of Ukraine", Depart of Neurinfections and Multiple Sclorosis, Kharkiv
  - Institue for Clinical Radiology of the State Establishment "Research Centre for Radiation Medicine of the AMS of Ukraino" Depart of Radiation Psychoneurology, Kiev
  - Vinnylsia Regional Psychoneurological Hosptial Named After O. I Yushchenko, Neurological Depart, Vinnytsia National Medical University Named After M. I. Pirogov, Chair of Neurology, Vinnitsa
- Rashid Hospital, Dubai, United Arab Emirates
- Kings College London, London, United Kingdom

REFERENCES:
- [Derived] Oh J, Walker B, Giovannoni G, Jack D, Dangond F, Nolting A, Aldridge J, Lebson LA, Leist TP. Side effects that occurred early in people with multiple sclerosis during the first year of treatment with cladribine tablets: a plain language summary. Neurodegener Dis Manag. 2022 Feb 1;12(1):1-7. doi: 10.2217/nmt-2021-0041. Epub 2022 Jan 12. PMID 35019731
- [Derived] Giovannoni G, Coyle PK, Vermersch P, Walker B, Aldridge J, Nolting A, Galazka A, Lemieux C, Leist TP. Integrated Lymphopenia Analysis in Younger and Older Patients With Multiple Sclerosis Treated With Cladribine Tablets. Front Immunol. 2021 Dec 24;12:763433. doi: 10.3389/fimmu.2021.763433. eCollection 2021. PMID 35003076
- [Derived] Giovannoni G, Galazka A, Schick R, Leist T, Comi G, Montalban X, Damian D, Dangond F, Cook S. Pregnancy Outcomes During the Clinical Development Program of Cladribine in Multiple Sclerosis: An Integrated Analysis of Safety. Drug Saf. 2020 Jul;43(7):635-643. doi: 10.1007/s40264-020-00948-x. PMID 32447743
- [Derived] Freedman MS, Leist TP, Comi G, Cree BA, Coyle PK, Hartung HP, Vermersch P, Damian D, Dangond F. The efficacy of cladribine tablets in CIS patients retrospectively assigned the diagnosis of MS using modern criteria: Results from the ORACLE-MS study. Mult Scler J Exp Transl Clin. 2017 Oct 9;3(4):2055217317732802. doi: 10.1177/2055217317732802. eCollection 2017 Oct-Dec. PMID 29051829
- [Derived] Leist TP, Comi G, Cree BA, Coyle PK, Freedman MS, Hartung HP, Vermersch P, Casset-Semanaz F, Scaramozza M; oral cladribine for early MS (ORACLE MS) Study Group. Effect of oral cladribine on time to conversion to clinically definite multiple sclerosis in patients with a first demyelinating event (ORACLE MS): a phase 3 randomised trial. Lancet Neurol. 2014 Mar;13(3):257-67. doi: 10.1016/S1474-4422(14)70005-5. Epub 2014 Feb 4. PMID 24502830
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=28821
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 617 participants were randomized for initial treatment period (ITP) and 616 participants received study drug.
Groups:
- Cladribine 5.25 mg/kg (ITP): Cladribine tablets administered as cumulative dose of 0.875 milligrams per kilograms (mg/kg) over a course of 5 consecutive days at Weeks 1, 5, 9, 13, 48, and 52 resulting in total cladribine dose of 5.25 mg/kg during the ITP of 96 weeks or until clinically definite multiple sclerosis (CDMS) conversion, whichever occurred first.
Period: ITP- Treatment Disposition
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP) | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Started | 205 | 206 | 206 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 204 | 206 | 206 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 104 | 131 | 104 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 101 | 75 | 102 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 20 | 10 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Converted to CDMS | 30 | 27 | 71 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 50 | 38 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: OLMP (Up to 96 Weeks)
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP) | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Started | 0 | 0 | 0 | 24 | 25 | 60 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 18 | 23 | 53 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 15 | 20 | 44 | 0 | 0 | 0 | 0 | 0 | 0
Period: LTFU (Cladribine Treatment) (48 Weeks)
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP) | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 17 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 17 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 16 | 0 | 0 | 0
Period: LTFU (No Cladribine) (48 Weeks)
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP) | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 36 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 36 | 14
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 36 | 14

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo).
Groups:
- Cladribine 5.25 mg/kg: Cladribine tablets administered as cumulative dose of 0.875 mg/kg over a course of 5 consecutive days at Weeks 1, 5, 9, 13, 48, and 52 resulting in total cladribine dose of 5.25 mg/kg during the ITP of 96 weeks or until CDMS conversion, whichever occurred first. Participants who converted to CDMS during ITP entered OLMP and received RNF subcutaneously at a dose of 44 mcg three times a week for up to 96 weeks. Participants who did not convert to CDMS during ITP, entered in LTFU period. Participants who converted to McDonald MS during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period.
- Cladribine 3.5 mg/kg: Cladribine tablets administered as cumulative dose of 0.875 mg/kg over a course of 5 consecutive days at Weeks 1, 5, 48, 52 and placebo matched to cladribine tablets was administered at Week 9 and 13 resulting in total cladribine dose of 3.5 mg/kg during the ITP of 96 weeks or until CDMS conversion, whichever occurred first. Participants who converted to CDMS during ITP entered OLMP and received RNF subcutaneously at a dose of 44 mcg three times a week for up to 96 weeks. Participants who did not convert to CDMS during ITP, entered in LTFU period. Participants who converted to McDonald MS during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any study treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period.
- Placebo: Placebo matched to cladribine tablets administered over a course of 5 consecutive days at Weeks 1, 5, 9, 13, 48 and 52 during the ITP of 96 weeks or until CDMS conversion, whichever occurred first. Participants who converted to CDMS during ITP entered OLMP and received RNF subcutaneously at a dose of 44 mcg three times a week for up to 96 weeks. Participants who did not convert to CDMS during ITP, entered in LTFU period. Participants who converted to McDonald MS during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period. Participants who did not convert to McDonald MS during ITP did not receive any study treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period.
- Total: Total of all reporting groups
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 204 | 206 | 206 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (8.8) | 31.7 (9.2) | 32.2 (8.2) | 31.9 (8.7)
Age, Customized [Count of Participants; unit: Participants]
  Greater than or equal to 30 years | 111 | 110 | 113 | 334
  Less than 30 years | 93 | 96 | 93 | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 130 | 138 | 400
  Male | 72 | 76 | 68 | 216
Expanded disability status scale (EDSS) score [Mean (Standard Deviation); unit: units on scale] — Expanded disability status scale (EDSS) assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
  units on scale | 1.6 (0.9) | 1.6 (0.9) | 1.7 (0.9) | 1.6 (0.9)
Number of Time Constant 1 (T1) Gadolinium Enhanced (GD+) lesions [Mean (Standard Deviation); unit: lesions] | 1.9 (5.8) | 1.5 (4.5) | 0.9 (2.5) | 1.4 (4.5)
Number of T2 Lesions [Mean (Standard Deviation); unit: lesions] | 29.7 (29.6) | 26.8 (28.3) | 26.3 (27.4) | 27.6 (28.4)
Time from First Demyelinating Event to Randomization [Mean (Standard Deviation); unit: Days] | 79.35 (17.61) | 78.67 (15.97) | 79.40 (17.94) | 79.14 (17.17)
Monofocal/Multifocal Classification (By Adjudication Committee) [Count of Participants; unit: Participants] — Monofocal- Neurological signs and symptoms can be explained by only 1 single location; Multifocal- Neurological signs and symptoms can not be explained by only 1 single location.
  Participants
    Monofocal | 108 | 112 | 101 | 321
    Multifocal | 96 | 94 | 105 | 295
Number of participants Using Steroid Treatment [Count of Participants; unit: Participants] | 133 | 131 | 140 | 404
Number of Participants with Time Constant 1 (T1) Gd-enhanced Lesions [Count of Participants; unit: Participants] | 90 | 74 | 73 | 237

OUTCOME MEASURES:

1. Primary Outcome: ITP: Time to Clinically Definite Multiple Sclerosis (CDMS) Conversion Represented by Kaplan-Meier Estimates of the Cumulative Percentage of Participants With CDMS
Description: CDMS according to the Poser criteria is defined as the occurrence of a second attack or a sustained increase in the expanded disability status scale (EDSS) Score. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to Multiple Sclerosis [MS]) was calculated. Sustained EDSS progression was defined as an increase in the EDSS score of greater than or equal to (>=) 1 point if baseline EDSS was between >= 1.0 and less than or equal to (=<) 4.5; or >= 1.5 points if baseline EDSS was 0, or >= 0.5 if baseline EDSS >= 5.0 over a period of at least 3 months. Kaplan-Meier estimates were provided for of the cumulative (cum.) percentage (%) of participants with CDMS over time. The probability of patients remaining event-free over time (from randomization) in each of the three treatment groups was displayed in the form of survival curves estimated using the non-parametric Kaplan-Meier method.
Time Frame: ITP: Baseline up to Week 96
Population: as for baseline characteristics
Measure: Number; unit: Cum. % of participants with CDMS
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Cum. % of participants with CDMS | 15.8 | 14.0 | 37.8
Statistical Analysis 1: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority or Other; p < 0.0001, two-sided Wald test — The treatment effect was also assessed by hazard ratios using the Cox's proportional hazards model; Hazard Ratio (HR) = 0.381, 95% CI 2-sided [0.248 to 0.584]
Statistical Analysis 2: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority or Other; p < 0.0001, two-sided Wald test — The treatment effect was also assessed by hazard ratios using the Cox's proportional hazards model; Hazard Ratio (HR) = 0.327, 95% CI 2-sided [0.210 to 0.509]

2. Secondary Outcome: ITP: Time to Develop Multiple Sclerosis (MS) Conversion According to the Revised McDonald Criteria (2005) Represented by Kaplan-Meier Estimates of the Cumulative Percentage of Participants With McDonald MS
Description: The McDonald criteria use dissemination in time and space established by magnetic resonance imaging (MRI) findings to provide a clinical diagnosis for MS. Dissemination in time is established by a new time constant 2 (T2) or gadolinium enhanced (Gd+) lesion found on a repeat MRI. Dissemination in space is established by the presence of any 3 of the following: 1 Gd+ lesion or 9 T2 bright lesions if there is no enhancement; greater than or equal to 1 infratentorial lesion; greater than or equal to 1 juxtacortical lesion; greater than or equal to 3 periventricular lesions. Kaplan-Meier estimates were provided for the cum. percentage (%) of participants with McDonald MS over time.
Time Frame: ITP: Baseline up to Week 96
Population: The ITT population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo).
Measure: Number; unit: Cum. % of participants with McDonald MS
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Cum. % of participants with McDonald MS | 51.36 | 56.05 | 87.14
Statistical Analysis 1: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority or Other; p < 0.0001, two-sided Wald test — The treatment effect was also assessed by hazard ratios using the Cox's proportional hazards model; Hazard Ratio (HR) = 0.425, 95% CI 2-sided [0.331 to 0.547]
Statistical Analysis 2: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority or Other; p < 0.0001, two-sided Wald test — The treatment effect was also assessed by hazard ratios using the Cox's proportional hazards model; Hazard Ratio (HR) = 0.497, 95% CI 2-sided [0.390 to 0.633]

3. Secondary Outcome: ITP: Number of Combined Unique Active (CUA) Lesions, New or Enlarging Time Constant 2 (T2) Lesions, and New or Persisting Time Constant 1 (T1) Gadolinium Enhanced (Gd+) Lesions Per Participant Per Scan
Description: Number of CUA lesions, new or enlarging T2 lesions, and new or persisting T1 Gd+ lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Baseline up to Week 96
Population: The ITT population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo). Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 203 | 202 | 196
Lesions
  CUA lesions | 1.20 (5.79) | 0.65 (1.80) | 2.13 (2.87)
  New or persisting T1 Gd+ lesions | 0.61 (5.33) | 0.29 (0.97) | 0.97 (1.62)
  New or enlarging T2 lesions | 0.62 (1.90) | 0.40 (1.12) | 1.17 (1.87)
Statistical Analysis 1: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); CUA lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.667, 95% CI 2-sided [-0.971 to -0.500]
Statistical Analysis 2: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); CUA lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.625, 95% CI 2-sided [-0.857 to -0.429]
Statistical Analysis 3: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); T1 Gd-Enhancing Lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.286, 95% CI 2-sided [-0.333 to -0.167]
Statistical Analysis 4: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); T1 Gd-Enhancing Lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.286, 95% CI 2-sided [-0.375 to -0.167]
Statistical Analysis 5: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); T2 Lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.333, 95% CI 2-sided [-0.500 to -0.167]
Statistical Analysis 6: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); T2 Lesions; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.286, 95% CI 2-sided [-0.429 to -0.143]

4. Secondary Outcome: OLMP: Time to 3 Month Confirmed Expanded Disability Status Scale (EDSS) Progression From Randomization Represented by Kaplan-Meier Estimates of Probability of Disability Progression
Description: EDSS progression is based on a standardized neurological exam and focuses on symptoms that commonly occur in Multiple Sclerosis (MS). Overall scores ranges from 0.0 (normal) to 10.0 (death due to MS). A sustained progression on EDSS score was defined as an EDSS progression confirmed into two consecutive assessment. Probability of disability progression at different time points was estimated using Kaplan-Meier method on the time to disability progression defined as the time from randomization to first EDSS increase.
Time Frame: OLMP: Day 1, 90, 180, 270, 360, 450, 540, 630, 720 and 810
Population: OLMP Analysis Set included all participants who received at least 1 dose of study medication, converted to CDMS in the ITP period, entered the OLMP and received at least 1 dose of OLMP study drug (Rebif). Here "Number analyzed" signifies those participants who were evaluable at specified time point for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Probability of Disability Progression
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 25 | 60
Probability of Disability Progression
  Day 1 | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]
  Day 90: number analyzed (Participants) | 24 | 24 | 59
  Day 90 | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]
  Day 180: number analyzed (Participants) | 22 | 21 | 52
  Day 180 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.0527 [-0.0054 to 0.1108]
  Day 270: number analyzed (Participants) | 21 | 18 | 47
  Day 270 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.0527 [-0.0054 to 0.1108]
  Day 360: number analyzed (Participants) | 18 | 14 | 40
  Day 360 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.0527 [-0.0054 to 0.1108]
  Day 450: number analyzed (Participants) | 12 | 10 | 30
  Day 450 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.0764 [0.0035 to 0.1492]
  Day 540: number analyzed (Participants) | 11 | 5 | 22
  Day 540 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.1094 [0.0147 to 0.2041]
  Day 630: number analyzed (Participants) | 7 | 3 | 13
  Day 630 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.1094 [0.0147 to 0.2041]
  Day 720: number analyzed (Participants) | 3 | 2 | 2
  Day 720 | 0.0417 [-0.0383 to 0.1216] | 0.0417 [-0.0383 to 0.1216] | 0.1094 [0.0147 to 0.2041]
  Day 810: number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Time to Conversion to Multiple Sclerosis (MS) According to the 2005 McDonald Criteria
Description: The McDonald criteria use dissemination in time and space established by magnetic resonance imaging (MRI) findings to provide a clinical diagnosis for MS. Dissemination in time is established by a new time constant 2 (T2) or gadolinium enhanced (Gd+) lesion found on a repeat MRI.
Time Frame: Time from Randomization up to 1217 days
Population: LTFU analysis set (No Treatment at LTFU Entry) consists of all participants who completed the 96-week ITP and entered the LTFU for safety follow-up and did not receive study treatment upon entry to the LTFU. Here "Number of Participants analyzed" signifies those participants who have been converted to CDMS.
Measure: Number; unit: Days
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 1 | 0 | 0
Days | 773 |  |

6. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) According to Poser Criteria
Description: CDMS according to the Poser criteria is defined as the occurrence of a second attack or a sustained increase in the expanded disability status scale (EDSS) Score. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. Sustained EDSS progression was defined as an increase in the EDSS score of greater than or equal to (>=) 1 point if baseline EDSS was between >= 1.0 and less than or equal to (=<) 4.5; or >= 1.5 points if baseline EDSS was 0, or >= 0.5 if baseline EDSS >= 5.0 over a period of at least 3 months.
Time Frame: Time from Randomization up to 1217 days
Population: LTFU analysis set (No Treatment at LTFU Entry) was used. Here "Number of Participants Analyzed" signifies those participants who have been converted to CDMS.
Measure: Number; unit: Days
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 1 | 0 | 0
Days | 773 |  |

7. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) According to Poser Criteria
Description: as for outcome 6
Time Frame: Time from Randomization up to 1217 days
Population: LTFU analysis set (Treated at LTFU Entry) analysis set consisted of all participants who converted to McDonald MS (2005) during the ITP, completed ITP 96-weeks and entered the LTFU. Here "Number of Participants analyzed" signifies those participants who have been converted to CDMS.
Measure: Number; unit: Days
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 0 | 0 | 1
Days |  |  | 767

8. Secondary Outcome: ITP: Percentage of Participants Converting to Clinically Definite Multiple Sclerosis (CDMS) as Per Poser Criteria
Description: Clinically definite multiple sclerosis (CDMS) according to the Poser criteria is defined as the occurrence of a second attack or a sustained increase in the expanded disability status scale (EDSS) Score. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. Sustained EDSS progression was defined as an increase in the EDSS score of greater than or equal to (>=) 1 point if baseline EDSS was between >= 1.0 and less than or equal to (=<) 4.5; or >= 1.5 points if baseline EDSS was 0, or >= 0.5 if baseline EDSS >= 5.0 over a period of at least 3 months. The percentage of participants who converted to CDMS are reported here.
Time Frame: ITP: Baseline up to week 96
Population: ITT analysis set included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Percentage of participants | 28.8 | 23.1 | 56.3

9. Secondary Outcome: ITP: Percentage of Participants Converting to McDonald Multiple Sclerosis (MS) (2005)
Description: Percentage of participants converting to mcDonald multiple sclerosis (2005) were reported.
Time Frame: ITP: Baseline up to week 96
Population: Intent-to-Treat analysis set included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Percentage of participants | 70.7 | 71.6 | 91.8

10. Secondary Outcome: ITP: Number of New or Persisting Gd-enhanced Lesions
Description: Number of new or persisting Gd-enhanced lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Week 13, 24, 36, 48, 60, 72, 84 and 96
Population: The intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo). Here "Number analyzed" signifies those participants who were evaluable at specified time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Lesions
  Week 13: number analyzed (Participants) | 188 | 189 | 192
  Week 13 | 0.86 (5.60) | 0.37 (1.52) | 1.00 (1.98)
  Week 24: number analyzed (Participants) | 171 | 186 | 166
  Week 24 | 0.03 (0.20) | 0.13 (0.51) | 0.92 (1.69)
  Week 36: number analyzed (Participants) | 105 | 115 | 100
  Week 36 | 0.08 (0.38) | 0.14 (0.44) | 0.74 (1.28)
  Week 48: number analyzed (Participants) | 163 | 173 | 143
  Week 48 | 0.02 (0.13) | 0.27 (0.92) | 0.87 (1.81)
  Week 60: number analyzed (Participants) | 145 | 148 | 131
  Week 60 | 0.10 (0.84) | 0.22 (0.94) | 0.74 (1.61)
  Week 72: number analyzed (Participants) | 128 | 146 | 115
  Week 72 | 0.05 (0.53) | 0.16 (0.81) | 0.90 (1.88)
  Week 84: number analyzed (Participants) | 116 | 126 | 83
  Week 84 | 0.02 (0.13) | 0.32 (2.62) | 0.60 (1.20)
  Week 96: number analyzed (Participants) | 70 | 80 | 49
  Week 96 | 0.07 (0.43) | 0.18 (0.84) | 0.64 (1.25)

11. Secondary Outcome: OLMP: Number of New or Persisting Gd-enhanced Lesions
Description: Number of new or persisting Gd-Enhanced lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 24, 48, 72 and 96
Population: OLMP Analysis Set included all participants who received at least 1 dose of study drug, converted to CDMS in ITP period, entered OLMP and received at least 1 dose of OLMP study drug. Here "Number of participants analyzed" = participants who were evaluable for this outcome measure and "Number analyzed" = who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 24 | 59
Lesions
  Baseline | 1.38 (5.52) | 0.88 (1.80) | 1.27 (2.58)
  Week 24: number analyzed (Participants) | 24 | 22 | 57
  Week 24 | 0.17 (0.48) | 0.05 (0.21) | 0.11 (0.56)
  Week 48: number analyzed (Participants) | 19 | 15 | 46
  Week 48 | 0.07 (0.24) | 0.00 (0.00) | 0.20 (0.50)
  Week 72: number analyzed (Participants) | 11 | 8 | 30
  Week 72 | 1.50 (3.28) | 0.13 (0.35) | 0.33 (1.18)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 1.58 (2.69) | 0.00 (0.00) | 0.07 (0.26)

12. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Number of New or Persisting Gd-enhanced Lesions
Description: Number of new or persisting Gd-Enhanced lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24 and 36
Population: LTFU analysis set (Treated at LTFU Entry) analysis set consisted of all participants who converted to McDonald MS (2005) during the ITP, completed ITP 96-weeks and entered the LTFU. Here "Number analyzed" signifies those participants who were evaluable at specified time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Lesions
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.71 (1.16)
  Week 13: number analyzed (Participants) | 7 | 8 | 16
  Week 13 | 0.00 (0.00) | 0.00 (0.00) | 0.13 (0.34)
  Week 24: number analyzed (Participants) | 7 | 8 | 11
  Week 24 | 0.00 (0.00) | 0.00 (0.00) | 0.18 (0.40)
  Week 36: number analyzed (Participants) | 2 | 3 | 10
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

13. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Number of New or Persisting Gd-enhanced Lesions
Description: Number of new or persisting Gd-Enhanced lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24, 36 and 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used. Here "Number analyzed" signifies those participants who were evaluable at specified time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Lesions
  Baseline | 0.00 (0.00) | 0.06 (0.23) | 0.14 (0.36)
  Week 13: number analyzed (Participants) | 22 | 23 | 11
  Week 13 | 0.00 (0.00) | 0.07 (0.23) | 0.09 (0.30)
  Week 24: number analyzed (Participants) | 15 | 15 | 5
  Week 24 | 0.00 (0.00) | 0.00 (0.00) | 0.20 (0.45)
  Week 36: number analyzed (Participants) | 4 | 7 | 3
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.17 (0.29)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 0.00 |  |

14. Secondary Outcome: ITP: Number of New or Enlarging T2 Lesions
Description: Number of new or enlarging T2 lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Week 13, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Lesions
  Week 13: number analyzed (Participants) | 188 | 189 | 192
  Week 13 | 1.56 (3.52) | 1.25 (3.33) | 1.43 (2.56)
  Week 24: number analyzed (Participants) | 171 | 186 | 166
  Week 24 | 0.24 (0.95) | 0.20 (0.66) | 1.01 (1.70)
  Week 36: number analyzed (Participants) | 104 | 115 | 100
  Week 36 | 0.09 (0.40) | 0.12 (0.42) | 1.14 (1.87)
  Week 48: number analyzed (Participants) | 165 | 174 | 143
  Week 48 | 0.07 (0.50) | 0.32 (2.52) | 1.04 (1.54)
  Week 60: number analyzed (Participants) | 145 | 148 | 131
  Week 60 | 0.13 (0.63) | 0.25 (1.09) | 0.71 (1.57)
  Week 72: number analyzed (Participants) | 128 | 148 | 116
  Week 72 | 0.03 (0.22) | 0.10 (0.34) | 0.83 (1.77)
  Week 84: number analyzed (Participants) | 116 | 127 | 83
  Week 84 | 0.09 (0.46) | 0.28 (2.03) | 0.61 (1.31)
  Week 96: number analyzed (Participants) | 69 | 79 | 50
  Week 96 | 0.04 (0.25) | 0.10 (0.59) | 0.38 (0.85)

15. Secondary Outcome: OLMP: Number of New or Enlarging T2 Lesions
Description: Number of new or enlarging T2 lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 24, 48, 72 and 96
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 24 | 60
Lesions
  Baseline | 0.29 (0.75) | 1.54 (6.72) | 2.13 (7.29)
  Week 24: number analyzed (Participants) | 23 | 22 | 57
  Week 24 | 0.26 (0.69) | 0.43 (1.35) | 0.68 (1.10)
  Week 48: number analyzed (Participants) | 19 | 16 | 46
  Week 48 | 0.32 (0.65) | 0.38 (1.09) | 0.41 (0.71)
  Week 72: number analyzed (Participants) | 11 | 8 | 30
  Week 72 | 0.95 (1.85) | 0.25 (0.46) | 0.97 (1.69)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 2.00 (3.52) | 0.67 (1.15) | 0.47 (1.06)

16. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Number of New or Enlarging T2 Lesions
Description: Number of new or enlarging T2 Lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Lesions
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.71 (1.53)
  Week 13: number analyzed (Participants) | 7 | 8 | 16
  Week 13 | 0.00 (0.00) | 0.25 (0.46) | 2.06 (4.25)
  Week 24: number analyzed (Participants) | 7 | 8 | 11
  Week 24 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Week 36: number analyzed (Participants) | 2 | 3 | 10
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.10 (0.32)

17. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Number of New or Enlarging T2 Lesions
Description: Number of new or enlarging T2 lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24, 36 and 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Lesions
  Baseline | 0.00 (0.00) | 0.03 (0.17) | 0.07 (0.27)
  Week 13: number analyzed (Participants) | 21 | 23 | 11
  Week 13 | 0.00 (0.00) | 0.04 (0.21) | 0.18 (0.40)
  Week 24: number analyzed (Participants) | 15 | 15 | 5
  Week 24 | 0.00 (0.00) | 0.13 (0.35) | 0.00 (0.00)
  Week 36: number analyzed (Participants) | 4 | 7 | 3
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.33 (0.58)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 0.00 |  |

18. Secondary Outcome: ITP: Number of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions
Description: Number of CUA lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Week 13, 24, 36, 48, 60, 72, 84 and 96
Population: ITT population included all randomized participants who received at least 1 dose of ITP study medication. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 189 | 189 | 192
Lesions
  Week 13 | 2.37 (6.87) | 1.56 (4.04) | 2.41 (3.89)
  Week 24: number analyzed (Participants) | 171 | 186 | 166
  Week 24 | 0.26 (1.03) | 0.29 (0.89) | 1.91 (2.93)
  Week 36: number analyzed (Participants) | 105 | 115 | 100
  Week 36 | 0.16 (0.71) | 0.25 (0.70) | 1.84 (2.64)
  Week 48: number analyzed (Participants) | 165 | 174 | 143
  Week 48 | 0.09 (0.59) | 0.56 (3.05) | 1.89 (2.78)
  Week 60: number analyzed (Participants) | 145 | 149 | 131
  Week 60 | 0.23 (1.40) | 0.42 (1.87) | 1.44 (2.70)
  Week 72: number analyzed (Participants) | 128 | 148 | 116
  Week 72 | 0.08 (0.72) | 0.22 (1.03) | 1.66 (3.05)
  Week 84: number analyzed (Participants) | 116 | 128 | 83
  Week 84 | 0.11 (0.51) | 0.55 (4.52) | 1.14 (1.95)
  Week 96: number analyzed (Participants) | 70 | 80 | 50
  Week 96 | 0.11 (0.60) | 0.23 (1.39) | 0.99 (1.89)

19. Secondary Outcome: OLMP: Number of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions
Description: Number of combined unique active (CUA) lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 24, 48, 72 and 96
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 24 | 60
Lesions
  Baseline | 0.63 (1.17) | 2.17 (7.72) | 3.23 (8.07)
  Week 24: number analyzed (Participants) | 24 | 22 | 57
  Week 24 | 0.42 (1.02) | 0.48 (1.40) | 0.79 (1.33)
  Week 48: number analyzed (Participants) | 19 | 16 | 46
  Week 48 | 0.39 (0.81) | 0.38 (1.09) | 0.61 (1.02)
  Week 72: number analyzed (Participants) | 11 | 8 | 30
  Week 72 | 2.45 (5.01) | 0.38 (0.74) | 1.30 (2.71)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 3.33 (6.03) | 0.67 (1.15) | 0.53 (1.25)

20. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Number of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions
Description: Number of CUA MRI lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24 and 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Lesions
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 1.24 (2.49)
  Week 13: number analyzed (Participants) | 7 | 8 | 16
  Week 13 | 0.00 (0.00) | 0.00 (0.00) | 2.19 (4.46)
  Week 24: number analyzed (Participants) | 7 | 8 | 11
  Week 24 | 0.00 (0.00) | 0.25 (0.46) | 0.18 (0.40)
  Week 36: number analyzed (Participants) | 2 | 3 | 10
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.10 (0.32)

21. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Number of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions
Description: Number of CUA lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24, 36 and 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Lesions
  Baseline | 0.00 (0.00) | 0.03 (0.17) | 0.14 (0.36)
  Week 13: number analyzed (Participants) | 22 | 23 | 11
  Week 13 | 0.00 (0.00) | 0.04 (0.21) | 0.18 (0.40)
  Week 24: number analyzed (Participants) | 15 | 15 | 5
  Week 24 | 0.00 (0.00) | 0.13 (0.35) | 0.00 (0.00)
  Week 36: number analyzed (Participants) | 4 | 7 | 3
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.33 (0.58)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 0.00 |  |

22. Secondary Outcome: ITP: Change From Baseline in Volume of T1 Gd-Enhanced Lesions
Description: Change in volume of T1 Gd-Enhanced lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Baseline, Week 96
Population: ITT population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo). Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm^3)
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 203 | 203 | 197
cubic millimeters (mm^3) | -73.97 (204.80) | -126.64 (399.39) | 48.63 (239.03)
Statistical Analysis 1: Comparison: Cladribine 3.5 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority; p < 0.0001, ANCOVA; Point Estimate = -1.700, 95% CI 2-sided [-37.200 to 0.000]
Statistical Analysis 2: Comparison: Cladribine 5.25 mg/kg (ITP) vs Placebo (ITP); Test type: Superiority; p < 0.0001, ANCOVA; Point Estimate = -28.600, 95% CI 2-sided [-117.300 to 0.000]

23. Secondary Outcome: OLMP: Mean Volume of T1 Gd-Enhanced Lesions and Changes From Baseline in Volume of T1 Gd-Enhanced Lesions
Description: Volume of T1 Gd-Enhanced lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 24, 48, 72 and 96
Population: OLMP Analysis Set was used. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 24 | 60
mm^3
  Baseline | 91.06 (368.98) | 113.64 (248.74) | 136.61 (344.31)
  Week 24: number analyzed (Participants) | 23 | 23 | 57
  Week 24 | 7.71 (26.35) | 3.48 (16.70) | 9.14 (55.62)
  Week 48: number analyzed (Participants) | 19 | 16 | 46
  Week 48 | 5.22 (19.75) | 0.00 (0.00) | 39.00 (188.80)
  Week 72: number analyzed (Participants) | 11 | 8 | 31
  Week 72 | 219.52 (377.85) | 56.86 (160.83) | 25.85 (96.18)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 330.20 (442.02) | 0.00 (0.00) | 22.51 (87.17)
  Change at Week 24: number analyzed (Participants) | 23 | 23 | 57
  Change at Week 24 | -87.30 (379.50) | -120.04 (250.42) | -134.67 (343.19)
  Change at Week 48: number analyzed (Participants) | 19 | 16 | 46
  Change at Week 48 | -106.82 (415.70) | -146.62 (298.86) | -116.06 (429.90)
  Change at Week 72: number analyzed (Participants) | 11 | 8 | 31
  Change at Week 72 | 26.00 (600.82) | -155.91 (341.97) | -192.24 (439.11)
  Change at Week 96: number analyzed (Participants) | 6 | 3 | 15
  Change at Week 96 | 275.83 (360.07) | -391.93 (523.92) | -247.76 (593.34)

24. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Mean Volume of T1 Gd-Enhanced Lesions and Changes From Baseline in Volume of T1 Gd-Enhanced Lesions
Description: Volume of T1 Gd-Enhanced lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24 and 36
Population: LTFU analysis set (Treated at LTFU Entry) was used. Here "Number analyzed" = participants evaluable at specified timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
mm^3
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 79.43 (143.64)
  Week 13: number analyzed (Participants) | 7 | 8 | 16
  Week 13 | 0.00 (0.00) | 0.00 (0.00) | 20.56 (70.96)
  Week 24: number analyzed (Participants) | 7 | 8 | 11
  Week 24 | 0.00 (0.00) | 0.00 (0.00) | 25.23 (66.24)
  Week 36: number analyzed (Participants) | 2 | 3 | 10
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Week 13: number analyzed (Participants) | 7 | 8 | 16
  Change at Week 13 | 0.00 (0.00) | 0.00 (0.00) | -63.83 (147.43)
  Change at Week 24: number analyzed (Participants) | 7 | 8 | 11
  Change at Week 24 | 0.00 (0.00) | 0.00 (0.00) | -32.25 (113.96)
  Change at Week 36: number analyzed (Participants) | 2 | 3 | 10
  Change at Week 36 | 0.00 (0.00) | 0.00 (0.00) | -58.93 (85.19)

25. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Mean Volume of T1 Gd-Enhanced Lesions and Changes From Baseline in Volume of T1 Gd-Enhanced Lesions
Description: Volume of T1 Gd-Enhanced lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 13, 24, 36 and 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used. Here "Number analyzed" = participants evaluable at specified timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
mm^3
  Baseline | 0.00 (0.00) | 4.45 (21.25) | 27.79 (76.02)
  Week 13: number analyzed (Participants) | 22 | 23 | 11
  Week 13 | 0.00 (0.00) | 7.34 (27.76) | 17.43 (57.80)
  Week 24: number analyzed (Participants) | 15 | 15 | 5
  Week 24 | 0.00 (0.00) | 0.00 (0.00) | 57.22 (127.95)
  Week 36: number analyzed (Participants) | 4 | 7 | 3
  Week 36 | 0.00 (0.00) | 0.00 (0.00) | 57.22 (99.10)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 0.00 |  |
  Change at Week 13: number analyzed (Participants) | 22 | 23 | 11
  Change at Week 13 | 0.00 (0.00) | 0.38 (1.32) | -17.95 (41.38)
  Change at Week 24: number analyzed (Participants) | 15 | 15 | 5
  Change at Week 24 | 0.00 (0.00) | -2.48 (9.60) | -20.60 (57.89)
  Change at Week 36: number analyzed (Participants) | 4 | 7 | 3
  Change at Week 36 | 0.00 (0.00) | -5.31 (14.06) | -31.48 (54.53)
  Change at Week 48: number analyzed (Participants) | 1 | 0 | 0
  Change at Week 48 | 0.00 |  |

26. Secondary Outcome: ITP: Changes From Baseline in Volume of T2 Lesions
Description: Change in volume of T2 lesions from baseline was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Baseline, Week 48 and 96
Population: ITT population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo). Here "Number analyzed" = participants evaluable at specified timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
mm^3
  Baseline | 3825.73 (5093.52) | 3435.22 (5184.12) | 3436.69 (4613.43)
  Change at Week 48: number analyzed (Participants) | 165 | 174 | 143
  Change at Week 48 | -654.20 (2061.85) | -828.97 (3513.04) | -29.57 (2581.44)
  Change at Week 96: number analyzed (Participants) | 70 | 81 | 51
  Change at Week 96 | -1237.44 (2718.76) | -1605.63 (2889.61) | -886.39 (2955.44)

27. Secondary Outcome: OLMP: Mean Volume of T2 Lesions and Changes From Baseline in Volume of T2 Lesions
Description: Volume of T2 lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 48 and 96
Population: OLMP Analysis Set was used. Here "Number analyzed" = participants evaluable at specified timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 25 | 60
mm^3
  Baseline | 398.88 (1102.27) | 630.70 (1707.24) | 1019.30 (2872.03)
  Week 48: number analyzed (Participants) | 19 | 16 | 47
  Week 48 | 767.66 (1875.86) | 458.13 (984.12) | 508.97 (1159.97)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 2606.15 (5542.81) | 0.00 (0.00) | 647.17 (1345.62)
  Change at Week 48: number analyzed (Participants) | 19 | 16 | 47
  Change at Week 48 | 523.27 (2065.54) | -20.20 (2025.21) | -77.67 (1760.20)
  Change at Week 96: number analyzed (Participants) | 6 | 3 | 15
  Change at Week 96 | 2245.18 (5810.53) | 0.00 (0.00) | 255.39 (1352.80)

28. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Mean Volume of T2 Lesions
Description: Volume of T2 lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline (Day 1)
Population: LTFU analysis set (Treated at LTFU Entry) was used.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
mm^3 | 1217.53 (1991.21) | 587.79 (1491.20) | 702.30 (1254.66)

29. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Mean Volume of T2 Lesions and Changes From Baseline in Volume of T2 Lesions
Description: Volume of T2 lesions was measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Baseline, Week 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used. Here "Number analyzed" = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
mm^3
  Baseline | 1402.08 (1799.96) | 962.26 (1026.99) | 1407.75 (1890.94)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 0.00 |  |
  Change at Week 48: number analyzed (Participants) | 1 | 0 | 0
  Change at Week 48 | -969.90 |  |

30. Secondary Outcome: ITP: Number of T1 Hypointense Lesions
Description: Number of T1 Hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: ITP: Baseline, Week 48 and 96
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Lesions
  Baseline | 8.0 (11.7) | 7.3 (12.2) | 7.0 (8.6)
  Week 48: number analyzed (Participants) | 162 | 171 | 141
  Week 48 | 8.39 (12.60) | 6.95 (12.86) | 7.07 (8.75)
  Week 96: number analyzed (Participants) | 69 | 79 | 48
  Week 96 | 5.35 (8.14) | 3.82 (6.89) | 5.06 (6.82)

31. Secondary Outcome: OLMP: Number of T1 Hypointense Lesions
Description: Number of T1 Hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: OLMP: Baseline, Week 48 and 96
Population: OLMP Analysis Set included all participants who received at least 1 dose of study medication, converted to CDMS in the ITP period, entered the OLMP and received at least 1 dose of OLMP study drug (Rebif). Here "Number analyzed" = participants evaluable at specified timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 25 | 60
Lesions
  Baseline | 0.92 (2.22) | 2.32 (9.52) | 1.45 (3.53)
  Week 48: number analyzed (Participants) | 19 | 15 | 46
  Week 48 | 3.79 (8.32) | 1.00 (2.85) | 0.74 (1.83)
  Week 96: number analyzed (Participants) | 6 | 3 | 15
  Week 96 | 0.50 (0.84) | 0.00 (0.00) | 1.47 (2.80)

32. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Number of T1 Hypointense Lesions
Description: Number of T1 Hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline (Day 1)
Population: LTFU analysis set (Treated at LTFU Entry) analysis set consisted of all participants who converted to McDonald MS (2005) during the ITP, completed ITP 96-weeks and entered the LTFU.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Lesions | 4.44 (7.25) | 1.22 (3.31) | 2.24 (5.01)

33. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Number of T1 Hypointense Lesions
Description: Number of T1 Hypointense lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: LTFU: Baseline, Week 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Lesions
  Baseline | 5.74 (8.21) | 3.53 (5.78) | 2.93 (4.46)
  Week 48: number analyzed (Participants) | 1 | 0 | 0
  Week 48 | 4.50 |  |

34. Secondary Outcome: ITP: Percentage of Participants With no New or Persisting T1 Gd-Enhanced Lesions
Description: T1 Gd-enhanced lesions were measured by using magnetic resonance imaging (MRI) scans. Percentage of participants with no new or persisting T1 Gd-enhanced lesions were reported.
Time Frame: ITP: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Percentage of Participants | 67.0 | 57.1 | 21.6

35. Secondary Outcome: OLMP: Percentage of Participants With no New or Persisting T1 Gd-Enhanced Lesions
Description: as for outcome 34
Time Frame: OLMP: Baseline up to Week 96
Population: OLMP Analysis Set included all participants who received at least 1 dose of study medication, converted to CDMS in the ITP period, entered the OLMP and received at least 1 dose of OLMP study drug (Rebif).
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 25 | 60
Percentage of participants | 25.0 | 50.0 | 35.3

36. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Percentage of Participants With no New or Persisting T1 Gd-Enhanced Lesions
Description: as for outcome 34
Time Frame: LTFU: Baseline up to Week 48
Population: LTFU analysis set (Treated at LTFU Entry) was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Percentage of Participants | 0 | 0 | 0

37. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Percentage of Participants With no New or Persisting T1 Gd-Enhanced Lesions
Description: as for outcome 34
Time Frame: Baseline up to Week 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Percentage of participants | 0 | 0 | 0

38. Secondary Outcome: ITP: Percentage of Participants With no New or Enlarging T2 Lesions
Description: T2 lesions were measured by using magnetic resonance imaging (MRI) scans. Percentage of participants with no new or enlarging T2 lesions were reported.
Time Frame: ITP: Baseline up to Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Percentage of Participants | 32.9 | 35.1 | 19.0

39. Secondary Outcome: OLMP: Percentage of Participants With no New or Enlarging T2 Lesions
Description: T2 Gd-enhanced lesions were measured by using magnetic resonance imaging (MRI) scans. Percentage of participants with no new or enlarging T2 Lesions were reported.
Time Frame: OLMP: Baseline up to 96
Population: as for outcome 35
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 24 | 25 | 60
Percentage of participants | 18.2 | 16.7 | 13.5

40. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Percentage of Participants With no New or Enlarging T2 Lesions
Description: Enlarging T2 Lesions were measured by using magnetic resonance imaging (MRI) scans. Percentage of participants with no New or Enlarging T2 Lesions were reported.
Time Frame: Baseline up to Week 48
Population: LTFU analysis set (Treated at LTFU Entry) was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Percentage of Participants | 0 | 0 | 0

41. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Percentage of Participants With no New or Enlarging T2 Lesions
Description: as for outcome 40
Time Frame: LTFU: Baseline up to Week 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Percentage of participants | 0 | 0 | 0

42. Secondary Outcome: ITP: Percent Change From Baseline in Brain Volume
Description: Brain volume was measured by using magnetic resonance imaging (MRI) scans. Percent change from baseline in brain volume at Week 48 and 96 was reported.
Time Frame: ITP: Baseline, Week 48 and 96
Population: The ITT population included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo). Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 155 | 163 | 135
Percent change
  Week 48 | -0.47 (0.63) | -0.48 (0.69) | -0.33 (0.76)
  Week 96: number analyzed (Participants) | 53 | 51 | 32
  Week 96 | -0.59 (0.80) | -0.72 (0.73) | -0.75 (0.65)

43. Secondary Outcome: OLMP: Percent Change From Baseline in Brain Volume
Description: as for outcome 42
Time Frame: OLMP: Baseline, Week 48 and 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP)
Number analyzed (Participants) | 5 | 4 | 11
Percent change
  Week 48 | -0.41 (0.98) | -1.60 (1.40) | -0.56 (1.11)
  Week 96: number analyzed (Participants) | 3 | 0 | 3
  Week 96 | 0.06 (1.36) |  | -1.31 (0.76)

44. Secondary Outcome: OLMP: Number of Relapses
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days.
Time Frame: Baseline up to Week 96
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 24 | 25 | 60
Relapses | 0.33 (0.64) | 0.16 (0.37) | 0.55 (1.00)

45. Secondary Outcome: LTFU (LTFU Analysis Set [Treated at LTFU Entry]): Number of Relapses
Description: as for outcome 44
Time Frame: Baseline up to Week 48
Population: LTFU analysis set (Treated at LTFU Entry) was used.
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU)
Number analyzed (Participants) | 9 | 9 | 17
Relapses | 0.00 (0.00) | 0.00 (0.00) | 0.06 (0.24)

46. Secondary Outcome: LTFU (LTFU Analysis Set [No Treatment at LTFU Entry]): Number of Relapses
Description: as for outcome 44
Time Frame: Baseline up to Week 48
Population: LTFU analysis set (No Treatment at LTFU Entry) was used.
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
Number analyzed (Participants) | 34 | 36 | 14
Relapses | 0.03 (0.17) | 0.03 (0.17) | 0.00 (0.00)

47. Secondary Outcome: OLMP: Annualized Relapse Rate
Description: The annualized relapse rate for each treatment group was the mean of the annualized relapse rates for all the participants in the group, calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25. Where, Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days.
Time Frame: Baseline up to Week 96
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 24 | 25 | 60
relapses per year | 0.24 [0.07 to 0.40] | 0.14 [0.00 to 0.27] | 0.42 [0.28 to 0.56]

48. Secondary Outcome: OLMP: Percentage of Relapse-Free Participants
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Percentage of relapse-free participants were reported.
Time Frame: Baseline up to Week 96
Population: OLMP Analysis Set included all participants who received at least 1 dose of study medication, converted to CDMS in the ITP period, entered the OLMP and received at least 1 dose of OLMP study drug (Rebif). Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 10 | 5 | 26
Percentage of participants | 40.0 | 20.0 | 30.8

49. Secondary Outcome: ITP: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. Number of Participants with TEAEs and serious TEAEs were reported.
Time Frame: ITP: Baseline up to Week 96
Population: Safety analysis set included all randomized participants who received at least 1 dose of ITP study medication (cladribine or placebo) and had at least one safety assessment during the ITP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP)
Number analyzed (Participants) | 204 | 206 | 206
Participants
  TEAEs | 165 | 168 | 162
  Serious TEAEs | 12 | 23 | 22

ADVERSE EVENTS:
Time Frame: ITP: Baseline up to 96 weeks; OLMP: Baseline up to 96 weeks; LTFU: Baseline up to 48 weeks
Description: ITP Safety analysis set(SAF). OLMP SAF: participants who received atleast 1dose of ITP study drug, converted to CDMS in ITP, entered OLMP and received atleast 1dose of OLMP study drug. LTFU (Treated)SAF: Participants who converted to McDonald MS(2005)during ITP, completed ITP 96-weeks and entered LTFU and treated with cladribine when entering LTFU. LTFU(Not-Treated) SAF:Participants who completed ITP 96-weeks and entered LTFU for safety follow-up and didn't receive study drug upon entry to LTFU.
Groups:
- Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU): Participants who received cladribine 5.25 mg/kg and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period . Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
- Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU): Participants who received cladribine 3.5 mg/kg and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period . Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
- Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU): Participants who received placebo and did not convert to CDMS during ITP, entered in long-term follow-up (LTFU) period. Participants who converted to McDonald multiple sclerosis (MS) during ITP or during LTFU period received open-label cladribine tablets (3.5 mg/kg) during LTFU period . Participants who did not convert to McDonald MS during ITP did not receive any treatment during LTFU period. Participants who converted to CDMS during LTFU received RNF subcutaneously at a dose of 44 mcg three times a week for the remaining LTFU period. Under the original study design, total duration of LTFU period was up to 96 weeks. The LTFU duration was reduced due to trial termination. Following the notice of trial termination, no further open label cladribine treatment was administered during the LTFU.
Arm/Group | Cladribine 5.25 mg/kg (ITP) | Cladribine 3.5 mg/kg (ITP) | Placebo (ITP) | Cladribine 5.25 mg/kg, Rebif (OLMP) | Cladribine 3.5 mg/kg, Rebif (OLMP) | Placebo, Rebif (OLMP) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) | Cladribine 5.25 mg/kg, Rebif (LTFU) | Cladribine 3.5 mg/kg, Rebif (LTFU) | Placebo, Rebif (LTFU)
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/206 | 0/206 | 0/24 | 1/25 | 0/60 | 0/9 | 0/9 | 0/16 | 0/34 | 0/36 | 0/14
Serious Adverse Events (participants affected / at risk) | 12/204 | 23/206 | 22/206 | 1/24 | 4/25 | 5/60 | 0/9 | 0/9 | 1/16 | 0/34 | 1/36 | 0/14
Other Adverse Events (participants affected / at risk) | 133/204 | 132/206 | 116/206 | 18/24 | 19/25 | 41/60 | 3/9 | 4/9 | 7/16 | 2/34 | 0/36 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 5.25 mg/kg (ITP) (N=204) | Cladribine 3.5 mg/kg (ITP) (N=206) | Placebo (ITP) (N=206) | Cladribine 5.25 mg/kg, Rebif (OLMP) (N=24) | Cladribine 3.5 mg/kg, Rebif (OLMP) (N=25) | Placebo, Rebif (OLMP) (N=60) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=9) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=9) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=16) | Cladribine 5.25 mg/kg, Rebif (LTFU) (N=34) | Cladribine 3.5 mg/kg, Rebif (LTFU) (N=36) | Placebo, Rebif (LTFU) (N=14)
Blood creatine phosphokinase increased (Investigations) | 3 | 7 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site necrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood amylase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillar neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 5.25 mg/kg (ITP) (N=204) | Cladribine 3.5 mg/kg (ITP) (N=206) | Placebo (ITP) (N=206) | Cladribine 5.25 mg/kg, Rebif (OLMP) (N=24) | Cladribine 3.5 mg/kg, Rebif (OLMP) (N=25) | Placebo, Rebif (OLMP) (N=60) | Cladribine 5.25 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=9) | Cladribine 3.5 mg/kg, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=9) | Placebo, Rebif, Cladribine 3.5 mg/kg (LTFU) (N=16) | Cladribine 5.25 mg/kg, Rebif (LTFU) (N=34) | Cladribine 3.5 mg/kg, Rebif (LTFU) (N=36) | Placebo, Rebif (LTFU) (N=14)
Lymphopenia (Blood and lymphatic system disorders) | 47 | 25 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 23 | 24 | 19 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 16 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 15 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 9 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 6 | 14 | 8 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 15 | 15 | 19 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 36 | 35 | 38 | 2 | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 21 | 17 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 14 | 21 | 13 | 2 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 12 | 10 | 12 | 2 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 17 | 13 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13 | 13 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 11 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 58 | 64 | 57 | 5 | 8 | 10 | 1 | 0 | 3 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 12 | 16 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 9 | 11 | 10 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 9 | 12 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 10 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 11 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 7 | 9 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radicular cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other